CLINICAL TRIAL: NCT03638284
Title: Non Invasive Brain Stimulation for Treatment of Neuropsychiatric Symptoms of Dementia: an Open Label Pilot Study Using Transcranial Direct Current Stimulation
Brief Title: Non-invasive Brain Stimulation Using Transcranial Direct Current Stimulation for Neuropsychiatric Symptoms of Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Sanjeev Kumar, Medical Head of Geriatric Clinical Research, Centre for Addiction and Mental Health; Clinician Scientist and Staff Psychiatrist, Campbell Family Mental Health Research Institute; Assistant Professor of Psychiatry, University of Toronto., Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 099/2017
Record Dates: First submitted 2018-07-13; First posted 2018-08-20 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Dementia; Alzheimer, Mixed Type (Etiology)
Keywords: Dementia; neuropsychiatric symptoms; tDCS; Transcranial direct current stimulation; Alzheimer Disease; Mixed Dementia; agitation in dementia; non-invasive brain stimulation
MeSH Terms: conditions — Dementia; Alzheimer Disease; Mixed Dementias; Aberrant Motor Behavior in Dementia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: All enrolled study participants will receive 10 sessions (5 per week X 2 weeks) of tDCS in an open label study. Participants will have neurocognitive assessments at baseline and at study completion (i.e. the last day of receiving tDCS).
Masking Description: N/a-open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transcranial Direct Current Stimulation (Experimental): Transcranial Direct Current Stimulation (tDCS):All enrolled study participants will receive 10 sessions (5 per week X 2 weeks) of tDCS in an open label study. Inhibitory stimulation will be delivered to the frontal lobes.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — tDCS is a non-invasive brain stimulation that does not require general anaesthesia or surgical implantation of a device. It uses two AA size batteries to deliver direct current via rubber electrodes enclosed in saline soaked sponges.

SUMMARY:
Agitation and aggression impose a tremendous burden on the individuals living with dementia, their families, caregivers, and healthcare systems. Neuropsychiatric symptoms of dementia (NPS) affect up to 80% of patients with Alzheimer's dementia. These symptoms impair patient and care giver's quality of life, increase the chances of hospitalization and also result in faster progression of the illness. The efficacy of current treatments is limited and the antipsychotic medications commonly used to treat these symptoms are associated with serious side effects. Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that uses a very low intensity electric current to modulate cortical excitability and brain plasticity. tDCS can be safely administered to awake persons and is very well tolerated. In this study the investigators will use tDCS to treat agitation related to NPSD.

DETAILED DESCRIPTION:
Agitation and aggression impose a tremendous burden on the individuals living with dementia, their families, caregivers, and healthcare systems. Neuropsychiatric symptoms of dementia (NPS) affect up to 80% of patients with Alzheimer's dementia. These symptoms include aggression and agitation, anxiety, depression, hallucinations, and delusions. These symptoms impair patient and care giver's quality of life, increase the chances of hospitalization and also result in faster progression of the illness. The efficacy of current treatments is limited and the antipsychotic medications commonly used to treat these symptoms are associated with serious side effects including cerebrovascular events, falls and increased risk of death. Electroconvulsive Therapy may be effective as well, however it requires anaesthesia and adversely affects cognition. Non-pharmacological or behavioral interventions are universally recognized as the first line treatment for agitation and NPSD. They are most effective when individualized and delivered in a person centered approach. Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that uses a very low intensity electric current to modulate cortical excitability and brain plasticity. tDCS can be safely administered to awake persons and is very well tolerated. Studies in healthy individuals and patients with Alzheimer's disease have shown that tDCS applied to frontal brain regions can enhance cognitive function. Further, tDCS applied to frontal brain regions can improve depressive symptoms. The effects of tDCS on NPSD are not known. In this study the investigators will use tDCS to treat agitation related to NPSD.The objective of this proposal is to conduct an open label pilot study of tDCS for treatment of agitation.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of Dementia of Alzheimer's, or Mixed type.
2. Presence of agitation and/or aggression related to NPS as defined by: Agitation in cognitive disorders; International Psychogeriatric Association Provisional Consensus Clinical and Research Definition at the time of enrolment into the study.
3. Patient or Substitute Decision Maker (SDM) able and willing to provide consent for enrolment in the study.
4. Age 60 or above

Exclusion Criteria:

1. Having dementia other than Alzheimer's or Vascular or Mixed type.
2. DSM-5 Axis I diagnoses other than dementia that is thought to be significantly impacting the presentation such as bipolar disorder, major depressive disorder, or schizophrenia
3. Imminent safety risk that would interfere with safe conduct of the study.
4. Any contraindication to tDCS such as metal implants in cranium.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
The rate of successful completion of the 2 week tDCS treatment course and rates of treatment associated adverse effects of tDCS in agitation due to NPSD | 2 weeks
  This will be assessed by the successful completion of the intervention in at least 80% of participants without any treatment associated serious adverse effects

SECONDARY OUTCOMES:
Effects of a 2 week course of tDCS on agitation as assessed by Cohen Mansfield Agitation Inventory (CMAI). | 2 weeks, 4 weeks
  Patients who undergo tDCS course will have reduced neuropsychiatric symptoms assessed using the Cohen Mansfield Agitation Inventory (CMAI). tDCS will result in a significant reduction in agitation as assessed by CMAI -frequency total score between baseline and post treatment follow up two weeks later. CMAI-frequency score ranges between 29 to 203 and CMAI-disruptiveness ranges from 29 to 145 for each category. Higher scores indicate worsening of symptoms.
Effects of a 2 week course of tDCS on agitation as assessed by Neuropsychiatric Inventory (NPI). | 2 weeks, 4 weeks
  Patients who undergo tDCS course will have reduced neuropsychiatric symptoms assessed using the Neuropsychiatric Inventory (NPI). tDCS will result in reduced burden of neuropsychiatric symptoms as assessed by Neuropsychiatric Inventory after the 2 week intervention. Each NPI domain is scored based on the interview conducted by the clinician. Frequency of symptoms are rated on a scale of 0 - 4 (Higher scores indicate symptoms occur more frequently). Severity / intensity of symptoms are rated on a scale of 0 to 3 (Higher scores indicate greater severity of symptoms). Caregiver distress is rated on a scale of 0 to 5 (Higher scores indicate increased caregiver distress).
Effects of a 2 week course of tDCS on agitation and other neuropsychiatric symptoms related to dementia as assessed by Clinical Global Impression (CGI). | 2 weeks, 4 weeks
  Patients who undergo tDCS course will have reduced neuropsychiatric symptoms as assessed using Clinical Global Impression -Improvement Scale CGI-I. tDCS will result in a significant improvement in clinical symptoms as assessed by CGI-I scale after the two week intervention. CGI-I scores range from 0-7, higher scores indicating worsening compared to at baseline.
Effect of tDCS on caregiver burden in agitation due to NPSD as assessed by Zarit Burden Interview (ZBI) | 2 weeks
  tDCS will result in significant reduction in caregiver burden as assessed by Zarit Burden Interview (ZBI). Scores on the ZBI range from 0 to 88, score of 0-21 indicating little or no burden; 21-40 indicating mild to moderate burden; 41-60 indicating moderate to severe burden; and 61-88 indicating severe burden.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Kumar, MD, FRCPC, Principal Investigator — CAMH
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No